CLINICAL TRIAL: NCT02479295
Title: Randomized Controlled Trial of Straight Versus Coiled Peritoneal Dialysis
Brief Title: Straight Versus Coiled Peritoneal Dialysis Catheter for Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chow Kai Ming, Dr, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015.197-T
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: End-stage Renal Disease; Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: straight versus coiled Tenckhoff catheters
Oversight: Data Monitoring Committee: No

ARMS (2):
- Straight Tenckhoff catheter (Active Comparator): Tenckhoff catheter with straight intra-abdominal part
  Interventions: Device: Tenckhoff catheter
- Coiled Tenckhoff catheter (Active Comparator): Tenckhoff catheter with coiled intra-abdominal part
  Interventions: Device: Tenckhoff catheter

INTERVENTIONS:
Device: Tenckhoff catheter — Peritoneal dialysis catheters for long term use
  Other Names: peritoneal dialysis catheter

SUMMARY:
This study compares the result of straight versus coiled Tenckhoff catheters for peritoneal dialysis patients. Recent meta-analysis of the peritoneal dialysis catheter type was in favor of straight catheters. The effects of straight versus coiled peritoneal dialysis catheters, however, are unclear. The investigators design an adequately powered randomized controlled study to evaluate the two types of double-cuffed peritoneal dialysis catheters. The primary objective is to assess whether straight peritoneal dialysis catheters can reduce the risk of catheter dysfunction that requires intervention. The investigators estimate that they would need to enroll 132 incident peritoneal dialysis patients in each group for the study to have 80% power to detect a difference between 7% and 15% in the primary endpoint of catheter dysfunction requiring intervention.

DETAILED DESCRIPTION:
The objective of the present study is to evaluate the a priori hypothesis that straight peritoneal dialysis catheters would improve the treatment outcomes of peritoneal dialysis. The early and late catheter complications, as well as catheter survival, will be compared between peritoneal dialysis patients who are randomized to straight and coiled Tenckhoff catheters.

ELIGIBILITY:
Inclusion Criteria:

* requires dialysis catheter insertion for maintenance peritoneal dialysis
* aged 18 or older
* willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* known contraindication to peritoneal dialysis
* participation in another interventional study within last 30 days of randomization
* history of a psychological illness or condition that would interfere with the patient's ability to understand the requirement of the study and/or comply with the dialysis procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of catheter dysfunction that requires intervention | One year
  Catheter dysfunction refers to drainage failure, as defined by the inability to drain peritoneal dialysate effluent reliably within 45 minutes. Intervention includes catheter repositioning or reinsertion, either by open surgical method or laparoscopically

SECONDARY OUTCOMES:
Time to catheter dysfunction requiring intervention | One year
  see above
Dialysis catheter migration with dysfunction | One year
  Dialysis catheter tip located above the pelvic brim on the abdominal radiograph
Infusion pain | One month
  Patient will be questioned on infusion pain around one month after starting peritoneal dialysis
Risk of peritonitis | One year
Technique failure | One year
Peritoneal dialysis catheter survival | One year

CONTACTS AND LOCATIONS:
Overall Officials: Kai Ming Chow, MBChB, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po

REFERENCES:
- [Derived] Chow KM, Wong SSM, Ng JKC, Cheng YL, Leung CB, Pang WF, Fung WWS, Szeto CC, Li PKT. Straight Versus Coiled Peritoneal Dialysis Catheters: A Randomized Controlled Trial. Am J Kidney Dis. 2020 Jan;75(1):39-44. doi: 10.1053/j.ajkd.2019.05.024. Epub 2019 Aug 21. PMID 31445925